CLINICAL TRIAL: NCT04835922
Title: Comparison of Efficacy of Intercostal Nerve Block vs Peritract Infiltration With 0.25% Bupivacaine in Percutaneous Nephrolithotomy: A Prospective Randomized Clinical Trial
Brief Title: Comparison of Efficacy of Intercostal Nerve Block vs Peritract Infiltration With 0.25% Bupivacaine in PCNL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Dr Sushil Gyawali, MS Resident, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 615-2020; REF/2021/01/000059 (Registry Identifier: NHRC trial registry number)
Record Dates: First submitted 2021-02-20; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Kidney Stone
Keywords: PCNL; Intercostal nerve block; Peritract Infiltration; Bupivacaine; Kidney stone
MeSH Terms: conditions — Kidney Calculi | interventions — Anesthesia, Conduction

STUDY DESIGN:
Intervention Model Description: the study will be prospective double blind randomized trial using 0.25% bupivacaine in patients undergoing PCNL under one of the two arms: Intercostal Nerve block or Peritract Infiltration.
Who Masked: Participant, Investigator
Masking Description: Double blinded study : participants and investigator will be blinded using sealed enveloped method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intercostal Nerve Block (Experimental): • In Group I (ICBN group): Intercostal nerve block will be given at 11th and 12th Intercostal space on the side of surgery with 20cc of 0.25% bupivacaine at the termination of PCNL under fluoroscopy guidance in prone position lateral to mid scapular line by Urologists. The 23 G spinal needle tip will be used and located above the innermost intercostal muscle. The needle tip will be located above the innermost intercostal muscle. In the next step, following negative aspiration for blood, 20 ml of 0.25% bupivacaine will be injected into the intercostal space between innermost intercostal muscle and pleura below 11th, and 12th ribs (10 ml each).
  Interventions: Procedure: Intercostal Nerve Block
- Peritract infiltration (Active Comparator): In Group P (PTI): Single dose of Peritract infiltration of 20cc of 0.25% bupivacaine will be given on completion of PCNL by Urologists. A 23 gauge spinal needle will be inserted up to the renal capsule along the nephrostomy tract at 6 and 12 o'clock (10ml at each position) under fluoroscopic guidance, 0.25 % bupivacaine will be infiltrated into the nephrostomy tract from renal capsule to the skin area (10 ml for each position). Then the surgical wound and intervention site will be covered with an occlusive dressing.
  Interventions: Procedure: Peritract Infiltration

INTERVENTIONS:
Procedure: Intercostal Nerve Block — : Following PCNL Intercostal nerve block will be given at 11th and 12th Intercostal space on the side of surgery with 20cc of 0.25% bupivacaine under fluoroscopy guidance in prone position lateral to mid scapular line by Urologists. The 23 G spinal needle tip will be used and located above the innermost intercostal muscle. The needle tip will be located above the innermost intercostal muscle. In the next step, following negative aspiration for blood, 20 ml of 0.25% bupivacaine will be injected into the intercostal space between innermost intercostal muscle and pleura below 11th, and 12th ribs (10 ml each)
  Other Names: Regional anesthesia
  Arms: Intercostal Nerve Block
Procedure: Peritract Infiltration — At the end of PCNL a single dose of Peritract infiltration of 20cc of 0.25% bupivacaine will be given by Urologists. A 23 gauge spinal needle will be inserted up to the renal capsule along the nephrostomy tract at 6 and 12 o'clock (10ml at each position) under fluoroscopic guidance, 0.25 % bupivacaine will be infiltrated into the nephrostomy tract from renal capsule to the skin area (10 ml for each position).
  Other Names: Regional anesthesia
  Arms: Peritract infiltration

SUMMARY:
Percutaneous nephrolithotomy (PCNL) is the preferred treatment for renal stones >2 cm or resistant to ESWL. Postoperative pain following this invasive surgery adds to the morbidity of patient which requires additional analgesia and can affect the quality of care. To lower the morbidity of PCNL, proper and adequate management of postoperative pain remains an integral component of PCNL.

There are many ways to reduce the postoperative pain following PCNL including mini PCNL, tubeless PCNL, use of regional analgesia etc. However the modality of analgesic technique is still a matter of debate. The aim of this study is to evaluate the efficacy of intercostal nerve block compared with peritract infiltration in patient undergoing PCNL. Specifically, the study will look on to the demography of patients undergoing PCNL and their indications. The study will also compare the intensity of pain in two groups using visual analogue scale (VAS). The study will be a prospective double blinded randomized clinical trial done at Department of Urology and Kidney Transplant Surgery, Tribhuvan University Teaching hospital (TUTH). The time frame of this study will be of 1 year or when sample size is fulfilled including all the patients who visit the hospital for PCNL and fulfils the inclusion criteria. At the end of our study we expect to conclude that the use of intercostal nerve block is superior or inferior than or equal to peritract infiltration in alleviating the postoperative pain following PCNL.

DETAILED DESCRIPTION:
Introduction:

The incidence and prevalence of renal calculi have increased globally across all ages, sex, and race, probably due to change in dietary habits and global warming. PCNL is considered 'gold standard' for the management of large renal calculi because it is less invasive and morbid than the open surgery. Currently, the indications for PCNL include large size renal calculi (>1.5-2 cm), staghorn calculi, upper tract calculi not responding to other modalities of treatment, lower pole stones, cystine nephrolithiasis, and stones in anatomically abnormal kidneys. However, the procedure causes postoperative pain, mostly due to dilatation of the renal capsule, the parenchyma and pain along the tract of the nephrostomy tube. So the postoperative pain remains an integral part of management. Postoperative pain management not only reduces patient suffering but also improve patient satisfaction, reduces morbidity and in parallel enhances recovery, improves rehabilitation, reduces hospital stay and thereby overall hospital cost. The postoperative pain due to the procedure may vary with individual pain perception, use of percutaneous nephrostomy (PCN) tubes, comorbid conditions, choice of analgesic route, anesthetic agents and postoperative course. Small calibers of tubes, even mini PCNL or tubeless PCNL and regional analgesia such as intercostal nerve block, peritract infiltration, paravertebral block etc. could further decrease postoperative pain and analgesic requirement and hence improving postoperative patient comfort. However, studies on these techniques have produced conflicting results due to the use of different local anesthetics, various regional techniques, and different study designs. So this study aims to compare the efficacy of intercostal nerve block and peritract infiltration with 0.25% bupivacaine in alleviating postoperative pain following the procedure with the subjective assessment of pain

Rational/justification :

• The optimal method of pain control after percutaneous nephrolithotomy remains controversial till now.

We need better technique of analgesia to decrease the pain following PCNL.

* Intercostal nerve block and peritract infiltration are common regional analgesic methods used by most of the investigators that had shown to be adequate for postoperative pain control.
* This study may be helpful in providing evidence for a clinical guideline to manage postoperative pain that will eventually help to decrease the morbidity and bring better outcome.

General Objective :

To compare the efficacy of intercostal nerve block and peritract infiltration with 0.25% bupivacaine in percutaneous nephrolithotomy.

Specific Objective :

* To analyse the demography of the patient [age, sex, BMI, stone size and laterality, renal function test, stone burden (size, Guy's Stone score etc.)] undergoing PCNL.
* To compare the intensity of pain using visual analogue score, resting and dynamic VAS scores, following PCNL between two groups (ICNB and PTI).
* To compare the time to first rescue analgesia and total analgesic requirement between both groups.
* To document the complications of both groups.

Research Hypothesis Is Intercostal nerve block more efficacious than peritract infiltration following PCNL in alleviating pain?

Study Variables

* Independent Variables: Age, Sex, BMI, stone location, laterality and size, Guys Stone score (burden), ASA grade, comorbidity, Group I (ICBN), Group P (PTI) nephrostomy tract size (mini vs standard), no of Tracts (single vs multiple), use to tube (tube vs tubeless), length of hospital stay, stone clearance, complications
* Dependent Variables R-VAS score, D-VAS score, Time to first analgesic demand, Total analgesic requirement

ELIGIBILITY:
Inclusion Criteria:

* All patients above 16 yrs of age undergoing PCNL in Tribhuvan University Teaching Hospital.

Exclusion Criteria:

* Patient ≤16 years of age, known history of hypersensitivity/anaphylaxis/ contraindications to bupivacaine, Systemic Diseases (CKD, active UTI, untreated sepsis), Relook surgery, high ASA grade ( >2) unfit for anesthesia/PCNL , Contraindications for PCNL (pregnancy, coagulopathy) , Patients who decline to participate

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-11-09 (Estimated); Study Completion 2021-11-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Score (VAS score) | up to 24 hours
  Patients undergoing PCNL who fulfil the inclusion criteria will be identified at the time of admission. • Patients will be randomized in two groups using sealed envelope method into ICNB (group I) and PTI (group P) prior to surgery. After the procedure (intervention) the intensity of pain will be evaluated by an independent observer (the researcher or an independent ward nurse) blinded to the allocated groups at postoperative 2, 8, 12 and 24 hours. The pain score will be assessed separately by Visual Analogue Scale (VAS), a 10-point scale ranging from 0, minimum or no pain, to 10, the maximum pain score perceived or imagined by the patient, at rest (RVAS) and on deep breathing or coughing known as dynamic VAS (DVAS). •

SECONDARY OUTCOMES:
Time to First Rescue analgesia | up to 24 hours
  Pain score will be recorded after the intervention as described earlier. Patients who will have VAS score of > 4 or intractable pain will be given rescue analgesia, that is injection ketorolac intravenously. The usual dose is 30 mg 4-6 hourly by the intravenous route. The time after procedure that patient needs first dose of rescue analgesia i.e Inj Ketorolac will be recorded. Dosage will be adjusted according to pain severity and response.
Total Analgesic Requiremennt | up to 24-48 hours
  Total Analgesia requirement of Inj Ketorolac required by the patient for the first 24 hours up to the discharge will be added up and recorded along with the time given.

CONTACTS AND LOCATIONS:
Overall Officials: Uttam Sharma, MS Surgery, Study Chair — HOD, Department of Urology and Kidney Transplant Surgery, TUTH
Locations (1):
- Tribhvan University Teaching Hospital, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No
After the research is completed, results will be published as Original Article in Journal. Relevant Individual data will be published in Journal itself as a part of the article.

REFERENCES:
- [Background] Jonnavithula N, Chirra RR, Pasupuleti SL, Devraj R, Sriramoju V, Pisapati MV. A comparison of the efficacy of intercostal nerve block and peritubal infiltration of ropivacaine for post-operative analgesia following percutaneous nephrolithotomy: A prospective randomised double-blind study. Indian J Anaesth. 2017 Aug;61(8):655-660. doi: 10.4103/ija.IJA_88_17. PMID 28890561
- [Background] Singh I, Yadav OK, Gupta S. Efficacy of intercostal nerve block with 0.25% bupivacaine in percutaneous nephrolithotomy: A prospective randomized clinical trial. Urol Ann. 2019 Oct-Dec;11(4):363-368. doi: 10.4103/UA.UA_141_18. PMID 31649454
- [Result] Choi SW, Cho SJ, Moon HW, Lee KW, Lee SH, Hong SH, Choi YS, Bae WJ, Ha US, Hong SH, Lee JY, Kim SW, Cho HJ. Effect of Intercostal Nerve Block and Nephrostomy Tract Infiltration With Ropivacaine on Postoperative Pain Control After Tubeless Percutaneous Nephrolithotomy: A Prospective, Randomized, and Case-controlled Trial. Urology. 2018 Apr;114:49-55. doi: 10.1016/j.urology.2017.12.004. Epub 2017 Dec 27. PMID 29288788
- See also: choi et al , Pubmed article, PCNL — https://pubmed.ncbi.nlm.nih.gov/29288788/